CLINICAL TRIAL: NCT01305525
Title: Partnership for Advancement In Neuromodulation (PAIN): A Prospective Clinical Outcomes Registry
Brief Title: A Prospective Clinical Outcomes Registry
Acronym: PAIN Registry
Status: Completed | Type: Observational
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Other Study IDs: C-09-01
Record Dates: First submitted 2011-02-25; First posted 2011-02-28 (Estimated); Last update posted 2019-01-30 (Actual); Status verified 2019-01

CONDITIONS: Pain
Keywords: SCS; St. Jude Medical; Neuromodulation
MeSH Terms: conditions — Pain

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Spinal Cord Stimulation
  Interventions: Device: St. Jude Medical Spinal Cord Stimulation Systems

INTERVENTIONS:
Device: St. Jude Medical Spinal Cord Stimulation Systems — Spinal cord stimulation

SUMMARY:
This is a prospective non-interventional 24 month post implant registry. Any patient that receives a St. Jude Medical FDA approved implantable neuromodulation system is eligible for enrollment. A minimum of 600 patients will be enrolled from a minimum of 30 sites.

Patients will be enrolled post-implant and followed for 24 months. Data are collected at enrollment (within 30 days of device implant), and routine care follow-up visits at 3 months, 6 months, 12 months, 18 months and 24 months.

ELIGIBILITY:
Inclusion Criteria:

1. Patient has signed and received a copy of the Informed Consent form;
2. Patient has been implanted with a St. Jude Medical Neuromodulation system, including battery and/or SCS leads;
3. Patient is 18 years of age or older.
4. Patient is not currently participating in another clinical trial.

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients implanted with a neuromodulation system
Sampling Method: Probability Sample
Enrollment: 614 (Actual)
Dates: Start 2009-06; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Patient reported outcomes over time | 2 years
  The primary objective of the registry is to create a prospective, outcome registry of patients implanted with neuromodulation devices.

CONTACTS AND LOCATIONS:
Locations (32):
- United States (31):
  - Scottsdale, Arizona
  - Azusa, California
  - Chula Vista, California
  - Sacramento, California
  - Jacksonville, Florida
  - Tampa, Florida
  - Evansville, Indiana
  - Muncie, Indiana
  - Louisville, Kentucky
  - Baton Rouge, Louisiana
  - Bloomfield Hills, Michigan
  - Waterford, Michigan
  - Saint Paul, Minnesota
  - Kalispell, Montana
  - New York, New York
  - Syracuse, New York
  - Utica, New York
  - Williamsville, New York
  - Durham, North Carolina
  - Winston-Salem, North Carolina
  - Mansfield, Ohio
  - Purcell, Oklahoma
  - Bethlehem, Pennsylvania
  - Houston, Texas
  - Southlake, Texas
  - Webster, Texas
  - Arlington, Virginia
  - Edmonds, Washington
  - Kirkland, Washington
  - Charleston, West Virginia
  - Morgantown, West Virginia
- San Juan, Puerto Rico